CLINICAL TRIAL: NCT04479397
Title: Post-operative Mobilization After Anterior Shoulder Stabilization With the Latarjet Procedure: Sling Versus Nothing. A Randomized Prospective Study.
Brief Title: Sling vs Nothing After Latarjet Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo Bothorel (Other)
Responsible Party: Sponsor-Investigator, Hugo Bothorel, Clinical trial supervisor LaTour Hospital, La Tour Hospital
Organization: La Tour Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-02469
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Shoulder Dislocation
Keywords: Latarjet; Post operative; Sling
MeSH Terms: conditions — Shoulder Dislocation | interventions — Postoperative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sling Arm (Active Comparator): This arm of the study will receive a sling for 3 weeks in postoperative care.
  Interventions: Procedure: Latarjet Surgery for anterior shoulder instability
- No Sling Arm (Experimental): This arm of the study will not receive a sling during the postoperative care,
  Interventions: Procedure: Latarjet Surgery for anterior shoulder instability; Procedure: No sling in postoperative care

INTERVENTIONS:
Procedure: Latarjet Surgery for anterior shoulder instability — Bone block procedure for anterior shoulder instability
Procedure: No sling in postoperative care — No sling will be used in postoperative care.
  Arms: No Sling Arm

SUMMARY:
Traumatic anterior shoulder instability is a common injury for the contact athlete, with high rates of recurrence in some athletic populations. The specific indication for the Latarjet procedure differs amongst surgeons, however it is generally accepted that it is indicated in patients with anterior glenohumeral instability that are unlikely to have a successful outcome from either an arthroscopic or open anatomical Bankart repair.

Overall the rate of reoperation following a Latarjet is around 5-7%. Infection, hematoma as well as screw removal and glenoid bony rim fractures are the most common indications for reoperation. The rate of instability after a Latarjet is low, with 1.7%-5.0% rate of dislocation.

However, in terms of rehabilitation, there are only a few studies and evidence of best practices. A recent review of the literature has highlighted four studies, comparing different rehabilitation protocols, which include different immobilization periods ranging from 0 to 3 weeks, and different types of mobilization (under physiotherapist supervision or not, with machine or not). They found a similar rate of recurrent dislocation between the different protocols. But early passive motion enables to improve the range of motion during first 3-6 months, with similar results at one year.

One main aspect which the surgeon can influence is immobilization time. In all above-mentioned studies, patients had to wear a sling for at least 3 weeks, even in the early mobilization groups. Short protocols with encouraging results have been recently emphasized by in other fields of shoulder surgery. The investigators would like to determine if the absence of postoperative immobilization could lead to improved function and better range of motion. To the investigators best knowledge, no study has sought to compare the usefulness of sling wearing after Latarjet procedure. Avoiding the sling could simplify rehabilitation and should provide a return to normal function faster.

DETAILED DESCRIPTION:
The aim of this study is to compare rehabilitation with the wearing of a sling, to rehabilitation without any immobilization after Latarjet procedure for treatment of anterior shoulder instability. Ultimately, the goal would be to offer to patients a simplified rehabilitation management, with a faster recovery, less pain and a quicker return to activities of daily living, work and sport.

As primary outcome, investigators will evaluate if the Rowe score is superior without postoperative immobilization (without a sling during the first 3 weeks) at 6 months after surgery compared to sling wearing.

Secondary outcomes include radiological criteria (X-rays and computed tomography (CT) at 6 months for bony union), return to sport, work absenteeism, other complication rate (especially redislocation), and the undermentioned subjective and clinical scores before surgery and at 1.5, 6 and 12 postoperative months.

All patients will be assessed with commonly used subjective scores in the form of self-administered questionnaires. The Visual Analog Scale (VAS) is a widely used single-item test where a patient rates pain intensity between 0 and 10. This scale is useful for patient preoperative and postoperative monitoring and has also been correlated with patient pain, anxiety and apprehension. Patient satisfaction (are patients satisfied, yes/no) will be assessed as well. Subjective Shoulder Value (SSV) is a single-question test where a patient is asked to rate his overall shoulder function as a percentage of normal shoulder. It is a quick and easily administered score that has also been validated for various shoulder disabilities, such as instability.

The following clinical scores will be analyzed as well Rowe score for instability is a three-item test with four choices each, measuring shoulder function, stability, and motion. The final result is converted into a value between 0 and 100. These scores have been specifically developed for shoulder instability.

Except for VAS, higher results mean higher function. ROM will be determined using a Vicon motion capture system (Vicon, Oxford Metrics, Oxford, UK) consisting of six cameras sampling at 120 Hz already available in our facility.

ELIGIBILITY:
Inclusion Criteria:

* all patients over 18 years old who have an anterior shoulder instability with one of the following criteria: an anterior glenoid bone defect > 20%, contact athlete or patients with failed Bankart repair-either open or arthroscopic will be considered eligible.

Exclusion Criteria:

* We exclude patients with a subscapularis tear, other trauma of the involved upper extremity (e.g. associated scapular or clavicular fractures, acromioclavicular dislocation), pre-operative stiffness, pre-operative sign of dislocation on standard X-ray, CT, CT arthrogram, MRI or MRA, contra-indication to CT (i.e pregnancy), and an inability to follow properly post-surgery recommendations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Rowe score | 12 postoperative months
  The Rowe Score consists of a total of 100 points divided into three domains: (1) stability, which corresponds to a total 50 points; (2) mobility, which corresponds to 20 points; (3) function, which corresponds to 30 points.

SECONDARY OUTCOMES:
The Visual Analog Scale (VAS) | 12 postoperative months
  The Visual Analog Scale (VAS) is a widely used single-item test where a patient rates pain intensity between 0 and 10. This scale is useful for patient preoperative and postoperative monitoring and has also been correlated with patient pain, anxiety and apprehension.
Subjective Shoulder Value (SSV) | 12 postoperative months
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percent- age of an entirely normal shoulder, which would score 100%.
Patient satisfaction | 12 postoperative months
  Patients will be asked "are you satisfied, yes/no"
Bony union | 12 postoperative months
  Will be evaluated using a CT scan and/or X-ray
Return to work | 12 postoperative months
  Time, in days, till patients return to work
Return to sport | 12 postoperative months
  Time, in days, untill patients return to sports
Redislocation | 12 postoperative months
  Did the shoulder redislocate postoperatively, yes or no
Range of motion | 12 postoperative months
  ROM will be determined using a Vicon motion capture system (Vicon, Oxford Metrics, Oxford, UK) consisting of six cameras sampling at 120 Hz already available in our facility.

CONTACTS AND LOCATIONS:
Locations (1):
- La Tour Hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Griesser MJ, Harris JD, McCoy BW, Hussain WM, Jones MH, Bishop JY, Miniaci A. Complications and re-operations after Bristow-Latarjet shoulder stabilization: a systematic review. J Shoulder Elbow Surg. 2013 Feb;22(2):286-92. doi: 10.1016/j.jse.2012.09.009. PMID 23352473
- [Result] Whitehouse T, Orr R, Fitzgerald E, Harries S, McLellan CP. The Epidemiology of Injuries in Australian Professional Rugby Union 2014 Super Rugby Competition. Orthop J Sports Med. 2016 Mar 22;4(3):2325967116634075. doi: 10.1177/2325967116634075. eCollection 2016 Mar. PMID 27069947
- [Result] van der Linde JA, van Wijngaarden R, Somford MP, van Deurzen DF, van den Bekerom MP. The Bristow-Latarjet procedure, a historical note on a technique in comeback. Knee Surg Sports Traumatol Arthrosc. 2016 Feb;24(2):470-8. doi: 10.1007/s00167-015-3704-7. Epub 2015 Aug 1. PMID 26231148
- [Result] An VV, Sivakumar BS, Phan K, Trantalis J. A systematic review and meta-analysis of clinical and patient-reported outcomes following two procedures for recurrent traumatic anterior instability of the shoulder: Latarjet procedure vs. Bankart repair. J Shoulder Elbow Surg. 2016 May;25(5):853-63. doi: 10.1016/j.jse.2015.11.001. Epub 2016 Jan 19. PMID 26809355
- [Result] Cunningham G, Ladermann A. Redefining anterior shoulder impingement: a literature review. Int Orthop. 2018 Feb;42(2):359-366. doi: 10.1007/s00264-017-3515-1. Epub 2017 Jun 6. PMID 28585076
- [Result] Ma R, Brimmo OA, Li X, Colbert L. Current Concepts in Rehabilitation for Traumatic Anterior Shoulder Instability. Curr Rev Musculoskelet Med. 2017 Dec;10(4):499-506. doi: 10.1007/s12178-017-9449-9. PMID 29038953
- [Result] Ialenti MN, Mulvihill JD, Feinstein M, Zhang AL, Feeley BT. Return to Play Following Shoulder Stabilization: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2017 Sep 14;5(9):2325967117726055. doi: 10.1177/2325967117726055. eCollection 2017 Sep. PMID 28944249
- [Result] Young AA, Maia R, Berhouet J, Walch G. Open Latarjet procedure for management of bone loss in anterior instability of the glenohumeral joint. J Shoulder Elbow Surg. 2011 Mar;20(2 Suppl):S61-9. doi: 10.1016/j.jse.2010.07.022. Epub 2010 Dec 9. No abstract available. PMID 21145262
- [Result] Ladermann A, Lubbeke A, Stern R, Cunningham G, Bellotti V, Gazielly DF. Risk factors for dislocation arthropathy after Latarjet procedure: a long-term study. Int Orthop. 2013 Jun;37(6):1093-8. doi: 10.1007/s00264-013-1848-y. Epub 2013 Mar 13. PMID 23508865
- [Result] Cunningham G, Benchouk S, Kherad O, Ladermann A. Comparison of arthroscopic and open Latarjet with a learning curve analysis. Knee Surg Sports Traumatol Arthrosc. 2016 Feb;24(2):540-5. doi: 10.1007/s00167-015-3910-3. Epub 2015 Dec 12. PMID 26658571
- [Result] Tirefort J, Schwitzguebel AJ, Collin P, Nowak A, Plomb-Holmes C, Ladermann A. Postoperative Mobilization After Superior Rotator Cuff Repair: Sling Versus No Sling: A Randomized Prospective Study. J Bone Joint Surg Am. 2019 Mar 20;101(6):494-503. doi: 10.2106/JBJS.18.00773. PMID 30893230
- [Result] Domos P, Lunini E, Ascione F, Serra N, Bercik MJ, Neyton L, Godeneche A, Walch G. Clinical and radiographic outcomes of open Latarjet procedure in patients aged 40 years or older. J Shoulder Elbow Surg. 2019 Sep;28(9):e304-e312. doi: 10.1016/j.jse.2019.02.004. Epub 2019 Apr 28. PMID 31043350
- [Result] Boileau P, Saliken D, Gendre P, Seeto BL, d'Ollonne T, Gonzalez JF, Bronsard N. Arthroscopic Latarjet: Suture-Button Fixation Is a Safe and Reliable Alternative to Screw Fixation. Arthroscopy. 2019 Apr;35(4):1050-1061. doi: 10.1016/j.arthro.2018.11.012. Epub 2019 Mar 8. PMID 30857907
- [Result] Gilbart MK, Gerber C. Comparison of the subjective shoulder value and the Constant score. J Shoulder Elbow Surg. 2007 Nov-Dec;16(6):717-21. doi: 10.1016/j.jse.2007.02.123. PMID 18061114
- [Result] Martinez-Urrutia A. Anxiety and pain in surgical patients. J Consult Clin Psychol. 1975 Aug;43(4):437-42. doi: 10.1037/h0076898. No abstract available. PMID 1159142
- [Result] Cunningham G, Zanchi D, Emmert K, Kopel R, Van De Ville D, Ladermann A, Haller S, Hoffmeyer P. Neural Correlates of Clinical Scores in Patients with Anterior Shoulder Apprehension. Med Sci Sports Exerc. 2015 Dec;47(12):2612-20. doi: 10.1249/MSS.0000000000000726. PMID 26110696
- [Result] Jensen KU, Bongaerts G, Bruhn R, Schneider S. Not all Rowe scores are the same! Which Rowe score do you use? J Shoulder Elbow Surg. 2009 Jul-Aug;18(4):511-4. doi: 10.1016/j.jse.2009.02.003. PMID 19559368
- [Result] Bessiere C, Trojani C, Pelegri C, Carles M, Boileau P. Coracoid bone block versus arthroscopic Bankart repair: a comparative paired study with 5-year follow-up. Orthop Traumatol Surg Res. 2013 Apr;99(2):123-30. doi: 10.1016/j.otsr.2012.12.010. Epub 2013 Mar 6. PMID 23481699
- [Result] Roulet S, Borel F, Franger G, Liotard JP, Michelet A, Godeneche A. Immediate self-rehabilitation after open Latarjet procedures enables recovery of preoperative shoulder mobility at 3 months. Knee Surg Sports Traumatol Arthrosc. 2019 Dec;27(12):3979-3988. doi: 10.1007/s00167-019-05635-8. Epub 2019 Jul 25. PMID 31346667
- [Result] Burkhart SS, De Beer JF, Barth JR, Cresswell T, Roberts C, Richards DP. Results of modified Latarjet reconstruction in patients with anteroinferior instability and significant bone loss. Arthroscopy. 2007 Oct;23(10):1033-41. doi: 10.1016/j.arthro.2007.08.009. PMID 17916467
- [Result] Park I, Oh MJ, Shin SJ. Minimal Clinically Important Differences and Correlating Factors for the Rowe Score and the American Shoulder and Elbow Surgeons Score After Arthroscopic Stabilization Surgery for Anterior Shoulder Instability. Arthroscopy. 2019 Jan;35(1):54-59. doi: 10.1016/j.arthro.2018.08.005. PMID 30611364
- [Derived] Goetti P, Martinho T, Seurot A, Bothorel H, Ladermann A. Is sling immobilization necessary after open Latarjet surgery for anterior shoulder instability? A randomized control trial. Trials. 2023 Feb 27;24(1):148. doi: 10.1186/s13063-023-07180-9. PMID 36850012